CLINICAL TRIAL: NCT00776243
Title: Short-term Effect of Intensive Insulin Therapy on Incretin Secretion
Status: Completed | Type: Observational
Sponsor: The Catholic University of Korea (Other)
Responsible Party: Kun-Ho Yoon, Kangnam St.Mary's hospital
Other Study IDs: KCMC08MI168; VCMC08OT066
Record Dates: First submitted 2008-10-20; First posted 2008-10-21 (Estimated); Last update posted 2010-05-12 (Estimated); Status verified 2009-10

CONDITIONS: Type 2 Diabetes
Keywords: incretin; GLP-1; GIP; intensive insulin therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma serum
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- wDM: Early diabetes
- pDM: Poorly controlled diabetic patients

SUMMARY:
In type 2 diabetic patients, abnormality in secretion or action of incretin(GLP-1, GIP) is observed. Although controversy still exists, the secretion of GLP-1 is thought to be reduced by 20-30% while GIP secretion is normal or slightly elevated, in type 2 diabetic patients. Various parameters such as the duration of diabetes, the amount of meal and their constitution, gastric bypass surgery, and some antidiabetic drugs affect the secretion of incretin. However, the secretion of GLP-1 and GIP in glucotoxic condition and whether they recover after improvement of glycemic status is not known. The investigators aim to study the effect of intensive insulin treatment in uncontrolled diabetic patients.

ELIGIBILITY:
Inclusion Criteria:

* type 2 diabetic patients with disease duration of less than 15years
* age of 20-70 years
* BMI 22-27
* HbA1c 9-13%
* patients willing to receive intensive glucose control
* patients who are able to monitor their glucose level at home

  * for normal glucose tolerance group : NGT subjects with same range of age and BMI
  * for early diabetes group : patients with diabetic duration of less than 5 years and HbA1c level less than 7.5% for at least last 6 months

Exclusion Criteria:

* previous history of insulin treatment
* patients taking alpha-glucosidase inhibitor or thiazolidinedione
* serum creatinine >= 1.5 mg/dL
* hemoglobin < 10 g/dL
* AST/ALT greater than 3 times normal range
* ischemic heart disease, congestive heart failure (NYHA grade >=2)
* chronic renal failure, proliferative diabetic retinopathy, CVA
* patients with gastroparesis or taking medications altering gastric motility
* usage of steroid or other agents affecting glucose metabolism
* pregnant or breast-feeding women

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Subjects with normal glucose tolerance
  2. Early diabetic patients with disease duration of less than 5years
  3. Uncontrolled diabetic patients
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2008-10; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Difference of incretin secretion before and after intensive insulin therapy | 2 months

SECONDARY OUTCOMES:
Difference in incretin secretion according to the duration of diabetes | basal
Factors affecting incretin secretion | basal

CONTACTS AND LOCATIONS:
Overall Officials: Kun-Ho Yoon, M.D., Ph.D., Principal Investigator — The Catholic University of Korea
Locations (2):
- South Korea (2):
  - Division of Endocrinology and Metabolism, St.Vincent's Hospital, Suwon, Kyonggi-do
  - Division of Endocrinology and Metabolism, Kangnam St.Mary's Hospital, Seoul

REFERENCES:
- [Background] Meier JJ, Nauck MA. Is secretion of glucagon-like peptide-1 reduced in type 2 diabetes mellitus? Nat Clin Pract Endocrinol Metab. 2008 Nov;4(11):606-7. doi: 10.1038/ncpendmet0946. Epub 2008 Aug 26. No abstract available. PMID 18725906
- [Background] Vollmer K, Holst JJ, Baller B, Ellrichmann M, Nauck MA, Schmidt WE, Meier JJ. Predictors of incretin concentrations in subjects with normal, impaired, and diabetic glucose tolerance. Diabetes. 2008 Mar;57(3):678-87. doi: 10.2337/db07-1124. Epub 2007 Dec 5. PMID 18057091
- [Background] Nauck MA, Baller B, Meier JJ. Gastric inhibitory polypeptide and glucagon-like peptide-1 in the pathogenesis of type 2 diabetes. Diabetes. 2004 Dec;53 Suppl 3:S190-6. doi: 10.2337/diabetes.53.suppl_3.s190. PMID 15561910
- [Background] Toft-Nielsen MB, Damholt MB, Madsbad S, Hilsted LM, Hughes TE, Michelsen BK, Holst JJ. Determinants of the impaired secretion of glucagon-like peptide-1 in type 2 diabetic patients. J Clin Endocrinol Metab. 2001 Aug;86(8):3717-23. doi: 10.1210/jcem.86.8.7750. PMID 11502801